CLINICAL TRIAL: NCT03866564
Title: The Football Players Health Study at Harvard University In Person Assessment Study
Brief Title: Football Players Health Study In Person Assessments Study
Acronym: IPA
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); Beth Israel Deaconess Medical Center (Other); Martinos Center for Biomedical Imaging (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Meagan Murphy Wasfy, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2018P001929
Record Dates: First submitted 2019-01-19; First posted 2019-03-07 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-03

CONDITIONS: Cardiac Dysfunction; Neurocognitive Disease; Chronic Pain; Sleep Apnea
MeSH Terms: conditions — Chronic Pain; Sleep Apnea Syndromes | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma & Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Multi-Afflicted: Participants with multiple self reported afflictions will undergo comprehensive research health screenings including Echocardiography (to define cardiac dysfunction), Neuropsychological Testing (to define neurocognitive disease), Pain Catastrophizing Scale (to define chronic pain), and Nocturnal Polysomnography (to define sleep apnea).
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Neuropsychological Testing; Diagnostic Test: Quantitative Sensory Testing; Diagnostic Test: Nocturnal Polysomnography
- Un-Afflicted: Participants who report no afflictions will undergo comprehensive research health screenings including Echocardiography (to define cardiac dysfunction), Neuropsychological Testing (to define neurocognitive disease), Pain Catastrophizing Scale (to define chronic pain), and Nocturnal Polysomnography (to define sleep apnea).
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Neuropsychological Testing; Diagnostic Test: Quantitative Sensory Testing; Diagnostic Test: Nocturnal Polysomnography
- Single Afflicted: Participants with one self reported afflictions will undergo comprehensive research health screenings including Echocardiography (to define cardiac dysfunction), Neuropsychological Testing (to define neurocognitive disease), Pain Catastrophizing Scale (to define chronic pain), and Nocturnal Polysomnography (to define sleep apnea).
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Neuropsychological Testing; Diagnostic Test: Quantitative Sensory Testing; Diagnostic Test: Nocturnal Polysomnography

INTERVENTIONS:
Diagnostic Test: Echocardiography — Cardiac ultrasound to measure left ventricular systolic function.
Diagnostic Test: Neuropsychological Testing — Standard clinical testing designed to establish or exclude the presence of cognitive dysfunction.
Diagnostic Test: Quantitative Sensory Testing — Clinically accepted quantitative assessment of chronic pain burden.
Diagnostic Test: Nocturnal Polysomnography — Routine overnight sleep study to measure apnea-hypopnea index.

SUMMARY:
The aim of the Football Players Health Study (FPHS) is to advance the understanding of the complex and inter-related pathways that can develop into player related illness and disability. Former National Football League players will be given the opportunity to undergo 2&1/2 days of rigorous assessment in the areas of Cardiac Dysfunction, Neurocognitive Disease, Chronic Pain, and Sleep Apnea to attempt to define the pathology among former professional athletes.

DETAILED DESCRIPTION:
Little is known about the long term health impacts of being exposed to a career in professional football. The primary objective of this study is to assess the relationship between affliction definitions, as subjectively described by participants in the first phase of the study (Q1), and objective pathology as defined by standard of care clinical and investigational testing. An exploratory secondary objective of this study is to examine the relationships between exposure to football, defined within the parameters of how old was the participant when their career started, how long did they play professional football, what was the participants field position and objective pathology defined as standard of clinical care.

The questions the study hopes to answer are as follows: 1) Are subjective complaints among former professional football players associated with objective evidence of pathology as measured by clinically accepted diagnostic testing (Primary objective), and 2) Is exposure to professional football, as defined by variables including career duration and player field position, associated with cardiac dysfunction, neurocognitive disease, chronic pain, and sleep apnea (Secondary objective).

This protocol has been constructed with an emphasis on reducing risk and maximizing yield. The Investigators who will be performing the assessments across the Harvard Medical School Institutions have worked together to minimize potential risk exposure by carefully selecting imaging protocols that limit radiation exposure, keeping phlebotomy limited, and by conducting these assessments under the supervision of investigators with established track records for conducting safe and effective human subject research.

The study visit will occur over 2&1/2 days. All costs of transportation, lodging, and meals will be covered by the study. All participants will have the assistance of a Study Navigator, a member of the FPHS staff who will accompany the participant. This navigator will assure that the participant gets to each assessment, helps to make decisions regarding scheduling issues or conflicts, assesses the need for additional breaks, and acts as a resource and guide for the participant throughout the study. The navigator will be in communication with key members of the research team for real time decision making (aborting or skipping an assessment).

Participants will be advised that results from these assessments are research results and are not meant for any diagnosis of disease. However, assessment results will be given to the participant if they wish to receive them. Any incidental finding that may have clinical relevance will be explained by a Study Physician and the Medical Navigation Nurse, and the participant will be assisted in obtaining follow up care.

ELIGIBILITY:
Inclusion Criteria:

* Age 24-55 at the time of first Health and Wellness Questionnaire (Q1) completion.
* Former professional football player who played between 1960 to present.
* Prior completed the first Health and Wellness Questionnaire (Q1)
* "Healthy" subjects: ability to give informed consent and comply with study procedures.
* "Afflicted" participants: must meet criteria for at least one of the following subjective afflictions based on Q1 responses: 1) Cardiovascular Dysfunction, 2) Neurocognitive Disease, 3) Chronic Pain, and/or 4) Sleep Apnea

Exclusion Criteria:

* Prior metallic device implants such as cardiac pacemakers/defibrillators or perfusion pumps that cannot be removed.
* Ferromagnetic implants or objects that cannot be removed such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants or jewelry
* Body weight >390 lbs at screening
* Inability to complete the telephone screener
* Low T-MoCA score (<17) and absence of an available study partner if required following MD review.
* Significant behavioral or functional disability due to cognitive impairment

Ages: 24 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women are not included in this study, as the National Football League is historically and currently a male-only entity
Study Population: Former Professional American-Style Football Players
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Cardiac Dysfunction | Study visit day 3
  Measurement of Left Ventricular Systolic Function (Ejection Fraction) by Transthoracic Echocardiography
Neurocognitive Disease | Study visit day 2
  Performance on Standard Clinical Neuropsychological Testing to Establish or Exclude Cognitive Impairment.
Chronic Pain: Pain Catastrophizing Scale | Study visit day 2
  Performance on Pain Catastrophizing Scale to Quantify the Magnitude of Chronic Pain. The range of this scale is from 0 to 52. The higher the score, the higher the presence of catastrophizing thoughts. A score of 30 or greater will be used to determine magnitude of pain that is clinically relevant
Sleep Apnea | study visit day 2
  Measurement of the Apnea-Hypopnea Index via Conventional Nocturnal Polysomnography. The Apnea-Hypopnea Index (AHI) is the measure of the number of apnea or hypopnea events measured in a one hour period. 0-5 events are normal, 6-15 events indicate mild sleep apnea, 16-30 events indicate moderate sleep apnea, over 30 events indicate sever sleep apnea. Scores of >15 will be considered positive for sleep apnea

CONTACTS AND LOCATIONS:
Overall Officials: Meagan M Wasfy, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States